CLINICAL TRIAL: NCT02200055
Title: The Use of Multifrequency Bioimpedance Assessments as an Estimate of Perioperative Total Body Volume and Postoperative Fluid Resuscitation
Brief Title: Using Electrical Bioimpedance Assessments to Estimate Perioperative Total Body Water and Postoperative Fluid Need
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Naval Medical Center, Portsmouth (U.S. Federal Agency)
Responsible Party: Principal Investigator, Christian McEvoy, General Surgery Resident, United States Naval Medical Center, Portsmouth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CIP# 12-0050
Record Dates: First submitted 2014-06-18; First posted 2014-07-25 (Estimated); Results first posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Intestinal Cancer; Diverticulitis; Pancreatic Cancer; Gastroesophageal Reflux Disease
Keywords: Electrical Bioimpedance; Major Intra-abdominal Surgical Procedures; Total Body Volume; Fluid Resuscitation
MeSH Terms: conditions — Intestinal Neoplasms; Diverticulitis; Pancreatic Neoplasms; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Bioimpedance Assessment (Experimental): The only group will be those patients having major intra-abdominal surgical procedures.
  Each patient involved in the study will be evaluated with a bioimpedance monitor ('Bodystat Quadscan 4000') to assess total body water, estimated body water, and intravascular body water volume preoperatively, postoperatively, and daily during the postoperative recovery period.
  Bioimpedance Assessment
  Interventions: Device: Bodystat Quadscan 4000

INTERVENTIONS:
Device: Bodystat Quadscan 4000 — Each patient involved in the study will be evaluated with a bioimpedance monitor to assess total body water, estimated body water, and intravascular body water volume preoperatively, postoperatively, and daily during the postoperative recovery period.
  Bioimpedance Assessment
  Other Names: Bioimpedance Assessment

SUMMARY:
Being able to accurately monitor patient bodily fluid levels during and after surgery is very important, as there are a number of complications that can arise if a patient's fluid levels become unbalanced, such as swelling within or pressure on various bodily organ systems. There are several different ways that physicians can monitor a patient's fluid balance during and after surgery, such as measuring the amount of urine output or the use of central venous catheters which measure the pressure in the veins entering the heart. Most of these techniques are invasive since they require tubes to be inserted into the body. A potential alternative would be to use a noninvasive technique such as electrical bioimpedance (BIA).

Bioimpedance assessments work by using small electrical currents that can accurately predict both the water surrounding the outside of cells in the body, as well as the total amount of water in the entire body. Electrical bioimpedance assessments have been used to estimate patient swelling following surgery (edema), to measure the volume of blood the heart is pumping out, as well as to calculate body fat percentages.

The goal of this study is to relate this technology to fluid shifts within the body that occur as a result of surgery, in particular, major intra-abdominal surgeries. By using bioimpedance during and after surgery, the investigators will compare the data collected with that calculated by using traditional measures of body fluid status, such as urine output and intraoperative blood loss. During the study, the bioimpedance monitors will not replace the standard bodily fluid monitors and will not interfere with their readings. Additionally, the electrical current produced by the bioimpedance monitors is too small for patients to feel and will not interfere with medical devices such as pacemakers.

DETAILED DESCRIPTION:
Being able to accurately monitor patient bodily fluid levels during and after surgery is very important, as there are a number of complications that can arise if a patient's fluid levels become unbalanced, such as swelling within or pressure on various bodily organ systems. There are several different ways that physicians can monitor a patient's fluid balance during and after surgery, such as measuring the amount of urine output or the use of central venous catheters which measure the pressure in the veins entering the heart. Most of these techniques are invasive since they require tubes to be inserted into the body. A potential alternative would be to use a noninvasive technique such as electrical bioimpedance (BIA).

Bioimpedance assessments work by using small electrical currents that can accurately predict both the water surrounding the outside of cells in the body, as well as the total amount of water in the entire body. Electrical bioimpedance assessments have been used to estimate patient swelling following surgery (edema), to measure the volume of blood the heart is pumping out, as well as to calculate body fat percentages.

The goal of this study is to relate this technology to fluid shifts within the body that occur as a result of surgery, in particular, major intra-abdominal surgeries. By using bioimpedance during and after surgery, the investigators will compare the data collected with that calculated by using traditional measures of body fluid status, such as urine output and intraoperative blood loss. During the study, the bioimpedance monitors will not replace the standard bodily fluid monitors and will not interfere with their readings. Additionally, the electrical current produced by the bioimpedance monitors is too small for patients to feel and will not interfere with medical devices such as pacemakers.

ELIGIBILITY:
Inclusion Criteria:

* Patients having major intra-abdominal procedures under general anesthesia requiring hospitalization postoperatively during the initial recovery from surgery.

Exclusion Criteria:

* Patients not having intra-abdominal procedures (ie. Thyroidectomy, open or laparoscopic inguinal hernia repair, excision of skin lesions, breast procedures)
* Patients having outpatient surgery
* Patients having laparoscopic cholecystectomies, laparoscopic or open appendectomies
* Patients having bariatric surgery (because the bioimpedance assessment technology has proven to be unreliable in obese populations)
* Morbidly obese patients (BMI >40)
* Unable to provide informed consent
* Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2012-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Oxner, MD, Principal Investigator — United States Naval Medical Center, Portsmouth
Locations (1):
- Naval Medical Center Portsmouth, Portsmouth, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Bioimpedance Assessment: The only group will be those patients having major intra-abdominal surgical procedures.
  Each patient involved in the study will be evaluated with a bioimpedance monitor to assess total body water, estimated body water, and intravascular body water volume preoperatively, postoperatively, and daily during the postoperative recovery period.
  Bioimpedance Assessment
  Bodystat Quadscan 4000: Each patient involved in the study will be evaluated with a bioimpedance monitor to assess total body water, estimated body water, and intravascular body water volume preoperatively, postoperatively, and daily during the postoperative recovery period.
  Bioimpedance Assessment
Period: Overall Study
Arm/Group | Bioimpedance Assessment
Started | 86
Completed | 86
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The number of participants meeting study eligibility requirements
Arm/Group | Bioimpedance Assessment
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 4
  Black or African American | 3
  White | 34
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Bioimpedance Assessment
Description: Bioimpedance assessment measurements were recorded for each participant before the surgical procedure
Time Frame: preoperative measurement
Population: This is the population of participants with bioimpedance measurements taken preoperative
Measure: Mean (Standard Deviation); unit: ohms
Groups:
- Bioimpedance Assessment: There are no groups for this study
Arm/Group | Bioimpedance Assessment
Number analyzed (Participants) | 45
ohms | 0.53 (0.06)

2. Primary Outcome: Bioimpedance Assessment
Description: Bioimpedance assessment measurements were recorded for each participant six hours following the surgical procedure
Time Frame: 6 hours postoperative measurement
Measure: Mean (Standard Deviation); unit: ohms
Groups:
- Bioimpedance Assessment: There are no groups in this study
Arm/Group | Bioimpedance Assessment
Number analyzed (Participants) | 45
ohms | 0.57 (0.07)

3. Primary Outcome: Bioimpedance Assessment
Description: Postoperative bioimpedance assessment measurements were recorded for each participant. One average across this time frame was recorded.
Time Frame: Average measurement, in ohms, taken daily for approximately 8-10 days
Population: This population of participants has their bioimpedance assessment taken daily for approximately 8-10 days postoperative. One average across this time frame was recorded
Measure: Mean (Standard Deviation); unit: ohms
Arm/Group | Bioimpedance Assessment
Number analyzed (Participants) | 45
ohms | 0.59 (0.24)

4. Secondary Outcome: Percent Extracellular Water Volume
Description: Extracellular water volume was recorded for each participant before surgical procedure.
Time Frame: preoperative measurement
Population: This is the final number of participants who met all study eligibility requirements
Measure: Mean (Standard Deviation); unit: percent of total water volume
Arm/Group | Bioimpedance Assessment
Number analyzed (Participants) | 45
percent of total water volume | 0.89 (3.68)

5. Secondary Outcome: Percent Intracellular Water Volume
Description: Intracellular water volume was recorded for each participant 6 hours following the surgical procedure.
Time Frame: 6 hour postoperative measurement
Measure: Mean (Standard Deviation); unit: percent of total water volume
Arm/Group | Bioimpedance Assessment
Number analyzed (Participants) | 45
percent of total water volume | 0.82 (1.54)

6. Secondary Outcome: Percent Extracellular Water Volume
Description: Extracellular water volume was recorded for each participant 6 hours following the surgical procedure.
Time Frame: 6 hours postoperative measurement
Population: This population contains data with extracellular water volume measurements taken post-operative
Measure: Mean (Standard Deviation); unit: percent of total water volume
Arm/Group | Bioimpedance Assessment
Number analyzed (Participants) | 45
percent of total water volume | 0.32 (0.34)

7. Secondary Outcome: Percent Intracellular Water Volume
Description: Intracellular water volume was recorded for each participant before surgical procedure.
Time Frame: Preoperative measurement
Population: This population includes data on participants with recorded intracellular water volume measurements
Measure: Mean (Standard Deviation); unit: percent of total water volume
Arm/Group | Bioimpedance Assessment
Number analyzed (Participants) | 45
percent of total water volume | 0.30 (0.04)
Statistical Analysis 1: Comparison: Bioimpedance Assessment; Test type: Superiority or Other — This measurement was collected for each participant. A pre-operative and post-operative bioimpedance measurement was taken; p < 0.01, Chi-squared; Mean Difference (Final Values) = 0.53

8. Secondary Outcome: Daily Fluid Balance (Intakes and Outputs)
Description: Each participant had a daily calculated fluid balance taken during the course of an approximate 8 day period
Time Frame: Sum of intakes and outputs each day while inpatient, an average of 8 days
Population: This was the final amount of participants who met all study eligibility requirements
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Bioimpedance Assessment
Number analyzed (Participants) | 45
mL | 1163.1 (1061.8)

9. Secondary Outcome: Urine Output
Description: Overall urine output was collected preoperative
Time Frame: preoperative measurement
Population: This population of participants recorded their urine output under preoperative conditions
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Bioimpedance Assessment
Number analyzed (Participants) | 45
mL | 406.7 (430.0)

10. Secondary Outcome: Study Characteristics of Participants: Body Mass Index
Description: Body Mass Index was recorded for each study participant at baseline
Time Frame: baseline measurement
Population: Baseline BMI was recorded for each participant
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Bioimpedance Assessment
Number analyzed (Participants) | 45
kg/m^2 | 27 (5)

11. Secondary Outcome: American Society of Anaesthesiologists Physical Status Classification Scale
Description: A classification scale to assess the fitness of patients before surgery
  The ASA score is a subjective assessment of a patient's overall physical health. The scale ranges from 1 to 5.
  ASA 1 A normal healthy patient. ASA 2 A patient with mild systemic disease. ASA 3 A patient with severe systemic disease. ASA 4 A patient with severe systemic disease that is a constant threat to life. ASA 5 A moribund patient who is not expected to survive
Time Frame: preoperative
Population: An ASA classification was recorded for each participant
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bioimpedance Assessment
Number analyzed (Participants) | 45
units on a scale | 2.2 (0.56)

12. Secondary Outcome: Amount of Intraoperative Fluids
Description: The amount of IV fluids each patient received during the surgical procedure
Time Frame: intraoperative measurement
Population: The population of participants with recorded data on the amount of IV fluids used during surgery
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Bioimpedance Assessment
Number analyzed (Participants) | 45
mL | 2472.6 (1147.0)

ADVERSE EVENTS:
Time Frame: Data collected April 2012 - 13November2014. Adverse event data were collected during that time and occurred between 19Aug2013 and 04Oct2014.
Description: At NMCP events are categorized as Adverse Events (AEs) or Serious Adverse Events (SAEs), depending on three criteria: Seriousness, expectedness, and relatedness to the research. An SAE must include all three criteria. SAEs are not limited to physical harms. They may include psychological, societal, and financial harms as well, such as psychological pain and embarrassment, loss of social standing, economic injury, loss of employment, potential for legal action, or loss of insurability, etc.
Arm/Group | Bioimpedance Assessment
All-Cause Mortality (participants affected / at risk) | 0/90
Serious Adverse Events (participants affected / at risk) | 3/90
Other Adverse Events (participants affected / at risk) | 3/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bioimpedance Assessment (N=90)
perineal wound infection (Infections and infestations) | 1 (1) — Post-op infection leading to hospital admission
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) — bronchospasm during surgery
upper gastrointestinal bleed (Gastrointestinal disorders) | 1 (1) — resulted in re-admission
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bioimpedance Assessment (N=90)
Pulmonary embolism (Vascular disorders) | 1 (1)
hemoperitoneum (Blood and lymphatic system disorders) | 1 (1)
pancreatic leak (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the number of participants who did not meet study eligibility requirements, we were only able to use 45 of 86 participants' data. Therefore, due such a small sample size, results from this study may lack generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes